CLINICAL TRIAL: NCT02320669
Title: Phase 3 Triiodothyronine Supplementation for Infants After Cardiopulmonary Bypass
Acronym: TRICC-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Responsible Party: Principal Investigator, Michael Portman, Principal Investigator, Seattle Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 14798; R01FD004362-01A2 (FDA)
Record Dates: First submitted 2014-12-05; First posted 2014-12-19 (Estimated); Results first posted 2024-04-09 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-03

CONDITIONS: Congenital Heart Defects
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Triiodothyronine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Triostat (Experimental): Active Medication - Synthetic Thyroid Hormone
  Interventions: Drug: Triostat
- Placebo (Placebo Comparator): Placebo Control
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Triostat — Bolus of Triiodothyronine followed by infusion for 48 hours
  Other Names: triiodothyronine
  Arms: Triostat
Drug: Placebo — Bolus of Placebo followed by infusion for 48 hours
  Arms: Placebo

SUMMARY:
This is a study to determine the safety and efficacy of liothyronine sodium/triiodothyronine (Triostat), a synthetic thyroid hormone, when given to infants with congenital heart disease during cardiopulmonary bypass surgery. Funding Source - FDA OOPD.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent obtained
2. Male and female patients <5 months (152 days) of age
3. Patients undergoing cardiopulmonary bypass

Exclusion Criteria:

1. Known thyroid disease (Down Syndrome is not an exclusion criterion unless patient has thyroid disease)
2. Trisomy 13 and 18
3. Prolonged preoperative ventilator support which would not be impacted by cardiac surgery (Lung disease: bronchopulmonary dysplasia, hypoplastic lungs associated with diaphragmatic hernia)
4. Any other condition as determined by the PI causing prolonged ventilator support which is unlikely to respond favorably to cardiac surgery
5. Prior participation in the clinical trial

Max Age: 5 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 220 (Actual)
Dates: Start 2014-11; Primary Completion 2019-10 (Actual); Study Completion 2019-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Portman, MD, Principal Investigator — Seattle Children's Hospital
Locations (3):
- United States (3):
  - Los Angeles Children's Hospital, Los Angeles, California
  - Lucille Packard Children's Hospital, Palo Alto, California
  - Seattle Children's Hospital, Seattle, Washington

REFERENCES:
- [Result] Portman MA, Slee AE, Roth SJ, Radman M, Olson AK, Mainwaring RD, Kamerkar A, Nuri M, Hastings L; TRICC Investigators. Triiodothyronine Supplementation in Infants Undergoing Cardiopulmonary Bypass: A Randomized Controlled Trial. Semin Thorac Cardiovasc Surg. 2023 Spring;35(1):105-112. doi: 10.1053/j.semtcvs.2022.01.005. Epub 2022 Jan 31. PMID 35093535

RESULTS

PARTICIPANT FLOW:
Groups:
- Triiodothyronine: Active Medication - Synthetic Thyroid Hormone Triostat: Bolus of Triiodothyronine followed by infusion for 48 hours
- Placebo: Placebo Control Placebo: Bolus of Placebo followed by infusion for 48 hours
Period: Overall Study
Arm/Group | Triiodothyronine | Placebo
Started | 110 | 110
Completed | 104 | 107
Not Completed | 6 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Triostat | Placebo | Total
Number analyzed (Participants) | 110 | 110 | 220
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 110 | 110 | 220
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: months] | 1.4 [.2 to 3.6] | 1.4 [0.2 to 3.6] | 1.4 [0.2 to 3.6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 41 | 84
  Male | 67 | 69 | 136
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 2 | 4
  Asian | 6 | 10 | 16
  Native Hawaiian or Other Pacific Islander | 2 | 2 | 4
  Black or African American | 2 | 5 | 7
  White | 71 | 62 | 133
  More than one race | 4 | 5 | 9
  Unknown or Not Reported | 23 | 24 | 47
Region of Enrollment [Number; unit: participants]
  United States | 110 | 110 | 220

OUTCOME MEASURES:

1. Primary Outcome: Time To Extubation
Description: time on mechanical ventilation after aortic cross clamp removal
Time Frame: 30 days
Population: modified intention to treat
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Triostat | Placebo
Number analyzed (Participants) | 110 | 110
hours | 46.9 [25.9 to 71.6] | 48.0 [31.0 to 65.4]
Statistical Analysis 1: Comparison: Triostat vs Placebo; Test type: Superiority; p < .05, Regression, Cox; Cox Proportional Hazard = 1.083, 95% CI 2-sided [.82 to 1.432]

2. Secondary Outcome: ICU Length of Stay
Description: Length of stay in the ICU
Time Frame: 30 days
Population: Children under age 5 mos undergoing cardiopulmonary bypass
Measure: Median (95% Confidence Interval); unit: days
Groups:
- Triiodothyronine: treatment group
- Placebo: Placebo group
Arm/Group | Triiodothyronine | Placebo
Number analyzed (Participants) | 110 | 110
days | 3.5 [2.3 to 4.8] | 2.9 [2.4 to 3.8]

ADVERSE EVENTS:
Time Frame: 30 days after receiving study medication
Description: Definitions were adopted from Pediatric Heart Network criteria
Arm/Group | Triostat | Placebo
All-Cause Mortality (participants affected / at risk) | 6/110 | 3/110
Serious Adverse Events (participants affected / at risk) | 11/110 | 11/110
Other Adverse Events (participants affected / at risk) | 17/110 | 20/110
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Triostat (N=110) | Placebo (N=110)
Sentinel (Cardiac disorders) | 11 (11) | 11 (11) — Sentinel including cardiac arrest and ECMO
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Triostat (N=110) | Placebo (N=110)
Cardiac Arrhythmia (Cardiac disorders) | 17 (110) | 20 (110) — Postoperative arrhythmia

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-09-30): https://cdn.clinicaltrials.gov/large-docs/69/NCT02320669/Prot_SAP_000.pdf